CLINICAL TRIAL: NCT00723424
Title: An Open-label Study to Assess the Effect of AZD5672 at Steady State on the Pharmacokinetics of Digoxin Following Single Dose Administration in Healthy Volunteers
Brief Title: Drug Interaction Study - Effect of AZD5672 on the Pharmacokinetics of Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Layton, MD, PhD, Medical Science Director, AstraZeneca R&D Alderely Park
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1710C00021; EudraCt nr 2007-007542-34
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers; Pharmacokinetics
Keywords: AZD5672; digoxin
MeSH Terms: interventions — N-(1-(3-(3,5-difluorophenyl)-3-(4-methanesulfonylphenyl)propyl)piperidin-4-yl)-N-ethyl-2-(4-methanesulfonylphenyl)acetamide; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD5672 + Digoxin (single dose on day 12)
  Interventions: Drug: AZD5672; Drug: Digoxin
- 2 (Experimental): AZD5672 (increasing dose up to 150mg) + digoxin (single dose on day 12)
  Interventions: Drug: AZD5672; Drug: Digoxin

INTERVENTIONS:
Drug: AZD5672 — 50 mg, for 13 days
Drug: Digoxin — 0.5mg dose
  Other Names: Lanoxin

SUMMARY:
The purpose of the study is to examine the effect of AZD5672 (dosed to steady state) on the pharmacokinetics of digoxin (single dose administration).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent.
* Females should not be of childbearing potential
* Clinically normal physical and laboratory findings as judged by the investigator, including negative drug test and negative tests of Hepatitis B surface antigen, antibodies to Hepatitis C virus and antibodies to HIV.

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subject's ability to participate
* Known allergy to digoxin or previous complications to digoxin therapy.
* Participation in any clinical study involving an investigational product in the 3 months prior to enrolment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during study periods

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Rod Hepburn, Study Director — AstraZeneca R&D, Charnwood, UK; Rainard Fuhr, Principal Investigator — Parexel
Locations (1):
- Research Site, Berlin, Germany